CLINICAL TRIAL: NCT05386264
Title: Production of Expanded Autologous Regulatory T Cells to Treat Patients With Refractory Aplastic Anaemia in a Phase I Dose Finding Study
Brief Title: Autologous Tregs for Aplastic Anaemia
Acronym: TIARA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-000082-33
Record Dates: First submitted 2022-02-18; First posted 2022-05-23 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Intervention Model Description: Open-label dose finding phase 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expanded autologous T regulatory cells (Experimental): This is an open-label, non-randomised interventional trial.
  Interventions: Other: Expanded autologous T regulatory cells

INTERVENTIONS:
Other: Expanded autologous T regulatory cells — A 3+3 dose escalation design with expanded T regulatory cells administered on Day 1 and Day 15

SUMMARY:
This Phase I study will determine the safety and optimal dose of expanded autologous Tregs to treat patients with Aplastic Anaemia (AA) (who have failed, or are considered ineligible for IST (immunosuppressive therapy) / other treatments) using expanded autologous T regulatory cells (Tregs) from AA patients at King's College Hospital, that have been prepared at the licensed Good Manufacturing Practices (GMP) production facility at Guy's Hospital, London

DETAILED DESCRIPTION:
The clinical trial will examine the safety of giving AA patients who have failed other treatment(s), their own ('autologous') expanded Tregs - a form of 'cellular therapy - to treat the AA. The investigators will study the changes in the immune system and determine if healthy bone marrow stem cells recover, thereby improving the blood counts after giving Tregs to patients. Expanded autologous Tregs are currently being looked at to treat other autoimmune disorders such as type I diabetes mellitus, multiple sclerosis, Crohn's disease and systemic lupus erythematosus. Results so far indicate that they are safe to give and do improve these diseases, but significantly this will be the first trial in AA.

ELIGIBILITY:
Inclusion Criteria:

* Acquired idiopathic AA
* No evidence of constitutional/inherited AA based on clinical findings, absence of family history of AA, normal DEB test and normal Kings bone marrow failure gene panel
* Very severe, severe or non-severe AA
* Lack a matched sibling donor (MSD) or matched unrelated donor (MUD), or ineligible for MSD/MUD HSCT
* Transfusion dependent
* Failed or ineligible for a course of ATG and CSA
* Failed / intolerant or inappropriate to treat with Eltrombopag or fails to meet Blueteq approval for use of Eltrombopag using NHS England guidance
* AST < 3 x upper limit of normal (ULN), bilirubin < 1.5 x ULN (unless Gilbert's syndrome)
* eGFR >50mL/min
* Age ≥ 18 years, male or female
* Willing and able to provide written and informed consent
* If female of child-bearing potential, have a negative serum pregnancy test and agree to use adequate contraceptive methods if of reproductive age
* Diffusing capacity for carbon monoxide (DLCO) ≥ 45% predicted corrected for haemoglobin
* LVEF > 40%.
* Performance status ≤ 2

Exclusion Criteria:

* Constitutional AA
* Age < 18 years' old
* Have a MSD and are eligible for MSD HSCT
* Have a MUD and are eligible for MUD HSCT
* Hypocellular myelodysplastic syndrome (Hypo MDS) or AA/Hypo MDS overlap
* Uncontrolled ongoing infection
* Active malignancy
* Treatment of cancer in the last 5 years (except in situ carcinoma of the cervix or basal cell carcinoma)
* Unable to give informed consent
* Active or uncontrolled infection not responding to appropriate antibiotics and antifungal agents.
* Human immunodeficiency virus (HIV) sero-positivity, hepatitis B, hepatitis C or hepatitis E infection.
* Abnormal organ function: AST/ALT >3 x upper limit of normal (ULN), bilirubin >1.5 x ULN, eGFR ≤50mL/min
* Heart failure (= grade III New York Heart Association)
* Pregnant or lactating women
* Unable or unwilling to comply with the contraceptive requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Expandability of functional T-regulatory cells from AA patients | Manufacturing to 24 months post final infusion
  This will be assessed through measuring the T regulatory cell count (1) during manufacturing production using a NC-200 cell counter and (2) through FACS analysis on peripheral blood research samples collected at the following 7 time points: pre-dose day 1, days 15, 29, 58 and at 6, 12 and 24 months
Assessment of safety and toxicity profile of the administrated autologous T-regulatory cells in AA patients | Baseline to 24 months post final infusion
  This will be assessed through physical examinations prior to each infusion and at every follow up visit. ECOG assessments prior to each infusions and at 6, 12 and 24 months. Bloods tests (FBC, Biochemistry, coagulation screen, d-dimer) prior to each infusion as well as 1 hour after infusion and 6 hours after the end of infusion). Bone marrow assessment prior to initial infusion and at 6, 12 and 24 months. AEs, SARs and SUSARs will be monitored from date of informed consent until 24 months. SAEs will be monitoring from date of informed consent until 30 days post final infusion. Adverse Events will be graded using CTCAE Version 5.0
Evaluation of safety and toxicity profile following 2 doses of autologous T-regulatory cells in AA patients | Baseline to 24 months post final infusion
  This will be assessed through physical examinations prior to each infusion and at every follow up visit. ECOG assessments prior to each infusions and at 6, 12 and 24 months. Bloods tests (FBC, Biochemistry, coagulation screen, d-dimer) prior to each infusion as well as 1 hour after infusion and 6 hours after the end of infusion). Bone marrow assessment prior to initial infusion and at 6, 12 and 24 months. AEs, SARs and SUSARs will be monitored from date of informed consent until 24 months. SAEs will be monitoring from date of informed consent until 30 days post final infusion. Adverse Events will be graded using CTCAE Version 5.0

SECONDARY OUTCOMES:
Response rate and duration of haematological response | Baseline to 24 months post final infusion
  This will be assessed by examining serial full blood counts, transfusion requirements and IV antibiotic usage on days D1, D2 D8, D15, D22, D29 and at 6, 12 and 24 months
Overall survival | 6 months to 24 months post final infusion
  Survival status will be determined by the trial clinician at 6, 12 and 24 months
Number and severity of infections | Baseline to 24 months post final infusion
  The number and severity of infections during first 30 days prior to starting Tregs will be compared to monthly average during therapy with Tregs until 24 months. This will be assessed through clinical examination and results of infection screening tests as recorded on EPR (Electronic Patient Records). Severity infections will be classified using the NCI Common Terminology Criteria for Adverse Events (CTCAE) for recording AEs and grade.
Clonal evolution to MDS/AML post treatment with Tregs | Baseline to 24 months post final infusion
  This will be assessed through (a) BM morphology (b) SNP-A karyotyping and (c) mutational profile, using Kings myeloid gene panel that includes 44 myeloid specific genes, at baseline (screening), 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Mufti, Study Director — King's College London
Locations (1):
- King's College Hospital, London, United Kingdom